CLINICAL TRIAL: NCT03391193
Title: Immunogenicity and Safety of a Multi-Dose Quadrivalent Influenza Vaccine in Children Aged 6 Months to 17 Years
Brief Title: Immunogenicity and Safety of a Multi-Dose Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GQM00016
Record Dates: First submitted 2017-12-21; First posted 2018-01-05 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent Inactivated Influenza Vaccine; Multi-dose Presentation
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-dose Quadrivalent Influenza Vaccine (Experimental): Quadrivalent influenza vaccine (split-virion, inactivated, 2017-2018 formulation, thiomersal containing) in multi-dose presentation. Participants aged 9 to 17 years will receive 1 dose and subjects aged 6 months to 8 years will receive 2 doses 28 days apart
  Interventions: Biological: Multi-dose Quadrivalent Influenza Vaccine
- Single-dose Quadrivalent Influenza Vaccine (Active Comparator): Quadrivalent influenza vaccine (split-virion, inactivated, 2017-2018 formulation, thiomersal free) in single-dose syringe presentation. Participants aged 9 to 17 years will receive 1 dose and subjects aged 6 months to 8 years will receive 2 doses 28 days apart
  Interventions: Biological: Single-dose Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Multi-dose Quadrivalent Influenza Vaccine — 0.5 mL, intramuscular
  Arms: Multi-dose Quadrivalent Influenza Vaccine
Biological: Single-dose Quadrivalent Influenza Vaccine — 0.5 mL, intramuscular
  Other Names: VaxigripTetra
  Arms: Single-dose Quadrivalent Influenza Vaccine

SUMMARY:
The aim of the study is to to assess the immunogenicity and safety of a quadrivalent influenza vaccine in a multi-dose presentation compared to a quadrivalent influenza vaccine in single-dose presentation, in children aged 6 months to 17 years.

DETAILED DESCRIPTION:
Participants aged 9 to 17 years will receive one dose of either the multi-dose quadrivalent influenza vaccine or the quadrivalent influenza vaccine in a single-dose presentation and participants aged 6 months to 8 years will receive 2 doses of either vaccine, 28 days apart.

All participants will provide a pre-vaccination blood sample on Day 0 and a post-vaccination blood sample either on Day 28 (participants aged 9 to 17 years) or on Day 56 (participants aged 6 months to 8 years) for immunogenicity testing.

All participants will be followed for safety evaluation up to 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 months to 17 years on the day of inclusion
* Assent form has been signed and dated by the subject aged 7 to 17 years, and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative and by an independent witness, if required by local regulations
* Subject and parent / legally acceptable representative are able to attend all scheduled visits and to comply with all study procedures
* Covered by health insurance, if required by local regulations

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche .
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, device, or medical procedure
* Receipt of any vaccine or planned receipt of any vaccine within the period from 2 weeks before the first study vaccination to 2 weeks following the last study vaccination
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccine or another vaccine for subjects aged 9 to 17 years.
* For subjects aged 6 months to 8 years:

  * Any influenza vaccination (from birth to the day of inclusion) with either the study vaccine or another vaccine
  * Any previous laboratory confirmed influenza infection
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Laboratory-confirmed / self-reported / reported by the parent(s) / legally acceptable representative Thrombocytopenia, contraindicating IM vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) of Antibodies after Vaccination with Multi-dose Quadrivalent Influenza Vaccine or Single-dose Quadrivalent Influenza Vaccine | Day 28 (post-last vaccination)
  Anti-hemagglutinin (HA) antibody titers against the 4 influenza strains are assessed by a hemagglutination inhibition (HAI) assay
GMT Ratio after Vaccination with Multi-dose Quadrivalent Influenza Vaccine or Single-dose Quadrivalent Influenza Vaccine | Day 28 (post-last vaccination)
  Anti-HA antibody titers against the 4 influenza strains are assessed by an HAI assay. GMT ratio is assessed as the individual ratio of post-/pre-vaccination titers
Seroconversion Rates after Vaccination with Multi-dose Quadrivalent Influenza Vaccine or Single-dose Quadrivalent Influenza Vaccine | Day 28 (post-last vaccination)
  Anti-HA antibody titers against the 4 influenza strains are assessed by an HAI assay. Seroconversion is defined as either post-vaccination titer ≥ 40 (1/dil), or pre-vaccination titer ≥ 10 (1/dil) and ≥ 4-fold increase in post-vaccination titer

SECONDARY OUTCOMES:
Percentage of Participants Reporting Solicited Injection Site or Systemic Reactions after Vaccination with Multi-dose Quadrivalent Influenza Vaccine or Single-dose Quadrivalent Influenza Vaccine | Day 0 (pre-vaccination) to Day 7 (after any vaccination)
  Solicited injection site reactions are tenderness/pain,erythema, swelling, induration, ecchymosis, and solicited systemic reactions are fever, vomiting, crying abnormal, drowsiness, appetite lost, irritability (for children ≤ 23 months), and fever, headache, malaise, myalgia, and shivering (for children 2 to 17 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- Mexico (3):
  - Sanofi Pasteur Investigational Site 0001, Cuernavaca, Morelos
  - Sanofi Pasteur Investigational Site 0002, Ecatepec de Morelos, State of Mexico
  - Sanofi Pasteur Investigational Site 0003, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org